CLINICAL TRIAL: NCT00321724
Title: A Phase II Trial of AZD2171 in Relapsed/Refractory B-Cell Chronic Lymphocytic Leukemia Patients
Brief Title: AZD2171 in Treating Patients With Relapsed or Refractory B-Cell Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01825; NCCTG-N048F; U10CA025224 (NIH); CDR0000467560 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2006-05-02; First posted 2006-05-04 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: B-cell Chronic Lymphocytic Leukemia; Refractory Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — cediranib

ARMS (1):
- Treatment (cediranib maleate) (Experimental): Patients receive oral AZD2171 once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cediranib maleate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: cediranib maleate — Given orally
  Other Names: AZD2171; Recentin
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well AZD2171 works in treating patients with relapsed or refractory B-cell chronic lymphocytic leukemia. AZD2171 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the cancer cells

DETAILED DESCRIPTION:
OBJECTIVES:

I. Evaluate the response rate in patients with relapsed or refractory B-cell chronic lymphocytic leukemia (B-CLL) treated with AZD2171.

II. Evaluate the toxicity of AZD2171 in patients with relapsed or refractory B-CLL.

III. Evaluate the complete response rate, progression-free and overall survival distributions, and duration of response in patients with relapsed or refractory B-CLL treated with AZD2171.

IV. Assess vascular endothelial growth factor receptor-2 (VEGFR-2) protein and phosphorylation levels in B-CLL cells using pretreatment samples and evaluate the association between Rai stage at study entry and clinical response to AZD2171.

V. Perform preclinical testing of AZD2171 in the induction of B-CLL cell apoptosis/cell death using pretreatment samples, and evaluate the ability to downregulate the phosphorylation status of VEGFR-2 of B-CLL cells by comparing in vitro samples with and without AZD2171.

VI. Study the differences in in vitro levels of B-CLL cell apoptosis/cell death and alteration of VEGFR-2 phosphorylation using pretreatment samples with and without AZD2171 and how these differences correlate with clinical outcomes.

VII. Assess if the clinical responses are associated with changes in bone marrow vascularity.

OUTLINE: This is a multicenter study.

Patients receive oral AZD2171 once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients undergo blood sampling and biopsies at baseline and periodically throughout study for biomarker and correlative studies.

After completion of study therapy, patients are followed periodically for up to 5 years from study entry.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of B-cell chronic lymphocytic leukemia (B-CLL)

  * Peripheral blood lymphocyte count > 5,000/mm³
  * Small to moderate peripheral blood lymphocytes with ≤ 55% prolymphocytes
  * Bone marrow aspirate with ≥ 30% lymphoid cells
  * Monoclonality of B lymphocytes by immunophenotyping, demonstrating all of the following:

    * B-cell markers with CD5 antigen in the absence of other pan-T-cell markers (CD3, CD2, etc.)
    * CD19 and/or CD20
    * Expression of CD23 on the CLL cells OR dim B-cell expression of kappa or lambda light chains
* Disease must be refractory to or progressive after treatment with at least 1 course containing a purine nucleoside analog (e.g., fludarabine, cladribine, or pentostatin)
* Life expectancy > 6 months
* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 50,000/mm³
* Hemoglobin ≥ 8 g/dL
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)

  * Patients with Gilbert's syndrome may have a bilirubin ≥ 1.5 times ULN
* AST and ALT ≤ 2.5 times ULN
* Creatinine ≤ 1.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of allergies to compounds similar to AZD2171
* QTc prolongation < 500 msec
* No other significant ECG abnormality
* No history of familial long QT syndrome
* Proteinuria < 1+ by dipstick OR protein < 1 g/24 hr urine collection
* No known HIV positivity
* No New York Heart Association (NYHA) class III or IV disease

  * NYHA class II disease controlled with treatment and monitoring allowed
* No other uncontrolled illness including, but not limited to, the following:

  * Hypertension
  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situations that would limit compliance
* See Disease Characteristics
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C), radiotherapy, anti-vascular endothelial growth factor (VEGF) treatment, or major surgery and recovered
* More than 30 days since prior investigational agents
* No concurrent drugs or biologics with proarrhythmic potential
* No other concurrent investigational agents
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2006-05; Primary Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Confirmed response defined to be an objective status of complete remission [CR], nodular partial remission [nPR], and partial remission [PR] | Up to 5 years
  Ninety percent confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner.

SECONDARY OUTCOMES:
Complete response rate estimated by the number of confirmed complete responses (CR) observed in the trial divided by the total number of evaluable patients | Up to 5 years
  Exact binomial 95% confidence intervals for the true complete response rate will be calculated.
Overall survival | From the date of registration to the date of death, assessed up to 5 years
  Estimated using the Kaplan-Meier method.
Time to progression as estimated by Kaplan-Meier method | From the date of registration to the date of disease progression, assessed up to 5 years
  Estimated using the Kaplan-Meier method.
Duration of response | From the date at which the patient's objective status is first noted to be a response to the date that progression or death is documented, assessed up to 5 years
  Estimated using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Kay, Principal Investigator — North Central Cancer Treatment Group
Locations (1):
- North Central Cancer Treatment Group, Rochester, Minnesota, United States